CLINICAL TRIAL: NCT05238857
Title: Investigation of Predisposing Factors Affecting Pain at Rest, During Activity, and at Night in Patients With Knee Osteoarthritis
Brief Title: Investigation of Predisposing Factors Affecting Pain in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University
Other Study IDs: 11012022
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Pain; Knee; Osteoarthritis; Function
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — There will be no intervention. Only assessments will be taken from the patients and data will be analyzed.

SUMMARY:
This study aims to determine the factors affecting pain in patients with knee osteoarthritis (OA). This study will be carried out following the "Helsinki Declaration", by selecting 106 volunteers who were diagnosed with knee OA, who applied to the Department of Orthopedics between February 2022 and August 2023 and met the inclusion criteria.

Before the evaluation, all the volunteers participating in the study will be informed about the purpose of the study, its duration, and the evaluations to be made. Consent will be obtained from all volunteers participating in the study with an "Informed Voluntary Consent Form". Demographic and clinical characteristics of all patients who voluntarily accepted to participate in the study will be questioned with the "Knee Osteoarthritis Evaluation Form". Quality of life, pain, range of motion (ROM), muscle strength, presence of comorbidity, and functional evaluation will be recorded on the form.

DETAILED DESCRIPTION:
Inclusion criteria:

- Volunteer participants who meet the clinical criteria for diagnosis of OA of the knee according to the American College of Rheumatology criteria will be included

Exclusion criteria:

* Diagnosis of neurologic disease, rheumatoid arthritis, radiculopathy or peripheral neuropathy, psychiatric disease
* History of knee surgery or intraarticular corticosteroid injection within the past 6 months
* Use of oral or topical analgesics for knee pain within the previous 6 months
* Receiving any physical therapy intervention on the lower limbs in the previous 6 months,
* Inability to read and write in Turkish
* Inability to follow simple instructions
* Having a pathology in visual ability and hearing

Assessments: Pain by Visual Analog Scale (VAS), ROM by digital goniometer, muscle strength by "Hand-held" dynamometer (Lafeyette Instrument®, Lafayette, IN), presence of comorbidity by Charlson Comorbidity Index, functional status WOMAC (Western Ontario and McMaster Universities) index, and quality of life will be evaluated with Short Form-12 (SF-12).

Statistics: The data obtained within the scope of the research will be analyzed with the Statistical Package for Social Science (IBM SPSS Statistics New York, USA) version 20.0. The distribution of the data will be evaluated with the "Shapiro Wilk Test". In the statistical analysis of the study, continuous variables will be shown with mean, standard deviation, minimum-maximum values, and categorical variables will be shown with frequency and percentage values. The relationship between VAS and independent factors will be analyzed with the "Pearson correlation test", and the effect of independent factors on the VAS score will be analyzed with "Linear Regression". In all analyses, p<0.05 (two-sided) values will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Volunteer participants who meet the clinical criteria for diagnosis of OA of the knee according to the American College of Rheumatology criteria will be included.

The exclusion criteria are as follows: (1) diagnosis of neurologic disease, rheumatoid arthritis, radiculopathy or peripheral neuropathy, psychiatric disease, (2) history of knee surgery or intraarticular corticosteroid injection within the past 6 months, (3) use of oral or topical analgesics for knee pain within the previous 6 months, (4) receiving any physical therapy intervention on the lower limbs in the previous 6 months, (5) inability to read and write in Turkish, (6) inability to follow simple instructions; and (7) having a pathology in visual ability and hearing.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All Females
Study Population: Women over the age of 40 years with knee osteoarthritis
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Baseline
  The pain severity will be assessed with Visual Analogue Scale (VAS), which is a numerical pain rating scale with zero corresponding to no pain and 10 corresponding to terrible pain.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline
  The health-quality of life of participants will be assessed with Short Form-12, which is a widely used reliable, valid, and responsive measure of quality of life in general population.
The Isometric Muscle Strength of Lower Extremity | Baseline
  The isometric strength of the iliopsoas, gluteus medius, quadriceps, and hamstring muscles of the affected side will be measured using a handheld dynamometer measuring kilogram per newton (Nicholas Manual Muscle Tester; model 01160, The Lafayette Instrument Company, Lafayette, Indiana). Each participant will be informed verbally about the technique of the test before starting. Each limb will assessed three times, with a 30-sec interval between tests, and the mean value will be calculated for analysis.
Functional Level of Lower Extremity | Baseline
  Functionality will be assessed with the Western Ontario and McMaster Universities Arthritis Index (WOMAC), which is a widely used reliable, valid, and responsive measure of outcome in people with osteoarthritis of the knee.
Active Range of Motion in Hip and Knee | Baseline
  The active range of motion, including hip flexion, knee flexion, and extension will be measured by using a digital goniometer (Baseline Evaluation Instrument, Fabrication Enterprises, Inc., White Plains, NY). Each participant will be informed verbally about the technique of the test before starting. The affected side will be assessed three times, with a 30-sec interval between tests, and the best value will be calculated for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No